CLINICAL TRIAL: NCT03098537
Title: Effects of Enteral Nutrition on Stress Ulcer Hemorrage. Multicenter Randomized Controlled
Brief Title: Effects of Enteral Nutrition on Stress Ulcer Hemorrage. Multicenter Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Kursat Gundogan, Associate Professor of Medicine and Surgery, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016/427
Record Dates: First submitted 2017-03-20; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Enteral Nutrition; Gastro Intestinal Bleeding; Stress Ulcer Prophylaxis; Proton Pump Inhibitor
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Enteral Nutrition; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral nutrion only (Active Comparator)
  Interventions: Other: enteral nutrition only
- Enteral nutrion + proton pump inhibitor (Other)
  Interventions: Drug: enteral nutrition + proton pump inhibitor

INTERVENTIONS:
Drug: enteral nutrition + proton pump inhibitor — Critically ill patients receiving any form of enteral nutrition will be included into the study. The patients will be randomized either enteral nutrition only group or enteral nutrition and proton pump inhibitors group. This group will receive enteral nutrition and proton pump inhibitor
  Arms: Enteral nutrion + proton pump inhibitor
Other: enteral nutrition only — Critically ill patients receiving any form of enteral nutrition will be included into the study. The patients will be randomized either enteral nutrition only group or enteral nutrition and proton pump inhibitors group. This group will receive only enteral nutrition.
  Arms: Enteral nutrion only

SUMMARY:
Enteral nutrition can provides prophylaxis against stress ulcer bleeding in critically ill patients and there may be no need to use acid suppressing drugs for stress ulcer bleeding prophylaxis in these patients. Half of the patients on enteral nutrition will not receive any acid suppressing drugs while other half receives it. They will be followed for gastrointestinal bleeding.

DETAILED DESCRIPTION:
Mucosal erosions can occur on luminal surface of stomach in approximately 75-100% patients during the first 24 hours of intensive care unit admission. These erosions often cause bleeding with penetrating superficial capillaries. Clinically significant bleeding (Significant decrease in blood pressure or decrease in hemoglobin level of more than 2 g / dL) appears to be less than 5% in ICU patients.

Enteral nutrition (EN) has protective effects against stress ulcer bleeding by neutralizing the acidic pH in the stomach lumen, providing a structural and functional integrity of the mucosal surface and trophic effect on the GI mucosa. These effects have been shown in some studies. The above-mentioned studies are inadequate for clinicians to make suggestions for relation between enteral nutrition and stress ulcer hemorrhage.

The risk factors for stress ulcer hemorrhage are mechanical ventilation, coagulopathy and burns.

Proton pump inhibitors (PPI) and histamine receptor blockers (H2RB) are the main drugs used for stress ulcer bleeding prophylaxis.

Studies have shown that 90% of patients admitted to intensive care units receive prophylaxis for stress ulcer bleeding.

Drugs (H2RB, PPI) used for prophylaxis against stress ulcer bleeding have some undesirable harmful effects in critical illnesses. These drugs, which suppress gastric acid secretion, can cause hospital-associated pneumonia and Clostridium difficile enterocolitis.

The studies, for clinical proposals are generally performed in the 1980s and early 1990s. Oral intake was stopped in most of the critically ill patients and early enteral nutrition was not widely used at the time of these major studies performed. Patients who are receiving EN have been shown to develop less stress ulcer bleeding in some studies. In a limited number of animal studies, enteral feeding has been shown to protect stress-related mucosal damage in the gastric mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Admission to ICU
* Expected to stay in ICU >24 hours
* No contraindications to EN within the first 24 hours after admission to the intensive care unit

Exclusion Criteria:

* Evidence of active GI bleeding during current hospitalization prior to study entry
* Coagulopathy (PLT<50.000, INR>1.5, aPTT>2xcontrol)
* Patients receiving acid suppressing drugs prior to admission
* Pregnancy or lactation
* History/documented gastric ulcer
* Burn>30% body surface area
* Head injury or increased intracranial pressure
* Partial or complete gastrectomy
* Shock
* Multi-system trauma
* Exposure to gastric irritant drugs
* Patients not giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
GI bleeding | Subjects will be followed from date of randomization until discharge from the ICU or cessation of enteral nutrition up to four weeks
  Overt GI bleeding (presence of coffee ground emesis hematemesis, melena or hematochezia.
  Significant GI bleeding, defined by 3-point decrease in hematocrit within 24 hours accompanied by overt GI bleeding or by an unexplained 6-point decrease in hematocrit during any 48 hour period.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Medical School, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook DJ, Fuller HD, Guyatt GH, Marshall JC, Leasa D, Hall R, Winton TL, Rutledge F, Todd TJ, Roy P, et al. Risk factors for gastrointestinal bleeding in critically ill patients. Canadian Critical Care Trials Group. N Engl J Med. 1994 Feb 10;330(6):377-81. doi: 10.1056/NEJM199402103300601. PMID 8284001
- [Background] Raff T, Germann G, Hartmann B. The value of early enteral nutrition in the prophylaxis of stress ulceration in the severely burned patient. Burns. 1997 Jun;23(4):313-8. doi: 10.1016/s0305-4179(97)89875-0. PMID 9248640
- [Background] Ephgrave KS, Kleiman-Wexler RL, Adair CG. Enteral nutrients prevent stress ulceration and increase intragastric volume. Crit Care Med. 1990 Jun;18(6):621-4. doi: 10.1097/00003246-199006000-00009. PMID 2111755
- [Background] Shorr LD, Sirinek KR, Page CP, Levine BA. The role of glucose in preventing stress gastric mucosal injury. J Surg Res. 1984 Apr;36(4):384-8. doi: 10.1016/0022-4804(84)90115-x. PMID 6546772
- [Background] Pingleton SK, Hadzima SK. Enteral alimentation and gastrointestinal bleeding in mechanically ventilated patients. Crit Care Med. 1983 Jan;11(1):13-6. doi: 10.1097/00003246-198301000-00005. PMID 6401236
- [Background] Cook DJ, Reeve BK, Guyatt GH, Heyland DK, Griffith LE, Buckingham L, Tryba M. Stress ulcer prophylaxis in critically ill patients. Resolving discordant meta-analyses. JAMA. 1996 Jan 24-31;275(4):308-14. PMID 8544272
- [Background] Daley RJ, Rebuck JA, Welage LS, Rogers FB. Prevention of stress ulceration: current trends in critical care. Crit Care Med. 2004 Oct;32(10):2008-13. doi: 10.1097/01.ccm.0000142398.73762.20. PMID 15483408
- [Background] Pisegna JR. Pharmacology of acid suppression in the hospital setting: focus on proton pump inhibition. Crit Care Med. 2002 Jun;30(6 Suppl):S356-61. doi: 10.1097/00003246-200206001-00003. PMID 12072661
- [Background] Lin PC, Chang CH, Hsu PI, Tseng PL, Huang YB. The efficacy and safety of proton pump inhibitors vs histamine-2 receptor antagonists for stress ulcer bleeding prophylaxis among critical care patients: a meta-analysis. Crit Care Med. 2010 Apr;38(4):1197-205. doi: 10.1097/CCM.0b013e3181d69ccf. PMID 20173630
- [Background] Herzig SJ, Howell MD, Ngo LH, Marcantonio ER. Acid-suppressive medication use and the risk for hospital-acquired pneumonia. JAMA. 2009 May 27;301(20):2120-8. doi: 10.1001/jama.2009.722. PMID 19470989
- [Background] Cunningham R, Dale B, Undy B, Gaunt N. Proton pump inhibitors as a risk factor for Clostridium difficile diarrhoea. J Hosp Infect. 2003 Jul;54(3):243-5. doi: 10.1016/s0195-6701(03)00088-4. PMID 12855243
- [Background] Dial S, Alrasadi K, Manoukian C, Huang A, Menzies D. Risk of Clostridium difficile diarrhea among hospital inpatients prescribed proton pump inhibitors: cohort and case-control studies. CMAJ. 2004 Jul 6;171(1):33-8. doi: 10.1503/cmaj.1040876. PMID 15238493